CLINICAL TRIAL: NCT01453231
Title: Quality of Life and Body Image in Women Underwent Thighplasty
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Ana Carolina Bim Tedesco, Physical Therapist, Federal University of São Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATedesco
Record Dates: First submitted 2011-10-13; First posted 2011-10-17 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Obesity
Keywords: bariatric surgery; plastic surgery; thigh; obesity; body image; quality of life
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): No surgery
- thighplasty (Experimental)
  Interventions: Procedure: thighplasty

INTERVENTIONS:
Procedure: thighplasty — Plastic surgery of thigh
  Arms: thighplasty

SUMMARY:
Obesity is a chronic disease now considered a major public health concern in the global context, as it causes or exacerbates many diseases limitations in providing quality of life and higher treatment costs. The increase in the number of patients undergoing bariatric surgery and the excess skin and subcutaneous tissue adjacent to slimming collaborate in the search for growth by plastic surgery. Currently several techniques of thighplasty has been submitted but no studies were found that evaluated the characteristic clinical and emotional resulting from this procedure. This study has as a goal to evaluate the body image and quality of life in women submitted to thighplasty.

DETAILED DESCRIPTION:
The patients have been evaluated for two different questionnaires, the Body Dysmorphic Disorder Examination (BDDE) and Impact Weight on Quality of Life - Lite (IWQoL-Lite). The sample consists of 50 patients with the desire to undergo to the thighplasty. However 25 are from study group and 25 control group. Just the study group was undergoing plastic surgery. The questionnaires have applied by signing the consent form, after 3 and 6 months both groups. This study is a clinical trial, control, primary, longitudinal, no random, analytical, held in a single center.

ELIGIBILITY:
Inclusion Criteria:

* abdominoplasty previous
* control of systemic disease
* Adults at the age of 35 and 50 years old
* had reached massive weight loss less by bariatric surgery or similar than 30 kg/m2 for a minimum of 12 months or more.
* gender: female
* For control group: it supposed to be on the waiting list for thighplasty
* For study group:they are supposed to be scheduled for thighplasty

Exclusion Criteria:

* illiterate
* pregnant women and/or women who have been nursing for one year or less
* non-controled of systemic disease

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-03; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
questionnaire about quality of life and body image | during 6 months
  The Questionnaires are apply three times, each 3 months, and until 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Tedesco, Master, Principal Investigator — Federal University of São Paulo
Locations (1):
- University Federal of Sao Paulo, São Paulo, São Paulo, Brazil